CLINICAL TRIAL: NCT00762541
Title: A Prospective Multicenter Trial To Evaluate The Safety And Effectiveness Of The MEL 80 Excimer Laser Using LASIK (Laser In Situ Keratomileusis) For The Correction Of > -7.00 D to -12.00 D Of Myopia With Up To -6.00 D Of Astigmatism, and Maximum MRSE of ≤ -12.00 D
Brief Title: Study of the MEL 80 Excimer Laser Using LASIK in the Treatment of Moderate to High Myopia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carl Zeiss Meditec, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MEL 80-2006-1
Record Dates: First submitted 2008-09-26; First posted 2008-09-30 (Estimated); Last update posted 2018-07-19 (Actual); Status verified 2018-07

CONDITIONS: Myopia
Keywords: Myopia; Laser In Situ Keratomileusis; Laser Therapy; Laser Corneal Surgery; Refractive Surgical Procedures; Ophthalmologic Surgical Procedure; Operative Surgical Procedures; Therapeutics
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: MEL 80 Treatment of High Myopia — The reduction or elimination of myopia > -7.00 D to -12.00 D, and astigmatism less than or equal to -6.00 D at the spectacle plane (myopia with or without astigmatism), with a maximum MRSE ≤ -12.00 D.

SUMMARY:
The purpose of this study is to determine whether the MEL 80 Excimer Laser is effective in the treatment of moderate to high myopia (nearsightedness), when used as part of the Laser In Situ Keratomileusis (LASIK) procedure.

DETAILED DESCRIPTION:
LASIK has become one of the most common refractive eye procedures performed in the country. Currently the MEL 80 Excimer Laser System is approved for the elimination of myopia of less than or equal to -7.0 D with or without refractive astigmatism of less than or equal to -3.0 D, with a maximum MRSE of -7.00 D. The goal of this study is to assess the safety and effectiveness information on the treatment of moderate to high magnitudes of myopia.

ELIGIBILITY:
Inclusion Criteria:

* Myopia > -7.00 D to -12.00 D, and astigmatism less than or equal to -6.00 D at the spectacle plane, with a maximum MRSE ≤-12.00 D.
* Stable refraction for at least the last twelve months, as demonstrated by a change of less than 1.00 D of the spherical equivalent during the twelve months prior to the baseline examination of the eye to be treated, documented by previous clinical records.
* Discontinue use of contact lenses at least 2 weeks for hard contacts and 3 days for soft lenses prior to the preoperative examination.
* Hard contact lens wearers must have two central keratometry readings and two manifest refractions taken at least one week apart that do not differ by more than 0.50 D.
* Visual acuity correctable to at least 20/40 in both eyes.
* UCVA of 20/40 or worse in the operative eye.
* At least 18 years of age.
* Operative eye must be targeted for emmetropia.
* Have a normal corneal topography.
* Willing and able to return for scheduled follow up examinations for twelve months after surgery.
* Sign and be given a copy of the written Informed Consent form.

Exclusion Criteria:

* History of anterior segment pathology, including cataracts (in the operative eye).
* Clinically significant dry eye syndrome unresolved by treatment.
* Residual, recurrent, active ocular or uncontrolled eyelid disease, corneal scars within the ablation zone or other corneal abnormality such as recurrent corneal erosion or severe basement membrane disease.
* Ophthalmoscopic signs of progressive or unstable myopia or keratoconus (or keratoconus suspect).
* An ablation deeper than 250 microns from the corneal endothelium.
* Irregular or unstable (distorted/not clear) corneal mires on central keratometry readings.
* Blind in the fellow eye.
* Undergone previous intraocular or corneal surgery of any kind in the operative eye(s), including any type of surgery for either refractive or therapeutic purposes.
* History of ocular Herpes zoster or Herpes simplex keratitis.
* History of steroid-responsive rise in intraocular pressure, glaucoma, or preoperative IOP >21 mm Hg.
* Must not have diabetes, diagnosed autoimmune disease, connective tissue disease, or clinically significant atopic syndrome.
* Must not be immunocompromised or use chronic systemic corticosteroid or other immunosuppressive therapy.
* Patients must not be pregnant, lactating, or of child-bearing potential and not practicing a medically approved method of birth control.
* Patients must not have a known sensitivity to planned study medications.
* Patients must not be participating in any other ophthalmic drug or device clinical trial during the time of this clinical investigation.
* For Fellow (Second) Eyes in Simultaneous Bilateral Treatment Procedures
* 1. Flap complications during the first eye's surgery such as a free cap, partial flap, thin flap, or irregular flap.
* 2. Epithelial defect exceeding 2 mm x 2 mm in dimension, or clinically significant debris in the interface between the flap and underlying stroma for the first eye.
* 3. Severe blepharospasm in the first eye that may have prevented or impeded the completion of the keratectomy and/or the laser ablation procedure.
* 4. Poor subject cooperation with instructions for the first eye's surgery and/or poor subject fixation on the laser fixation target.
* 5. Aborted LASIK procedure in the first eye or PRK was performed in the first eye because LASIK was not possible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2006-10; Primary Completion 2008-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
At the point of stability, for myopes > 7 D spherical equivalent (SE), a minimum of 30% should have an achieved refraction within ± 0.50 D of the intended outcome, and 60% should have an achieved refraction within ± 1.00 D of the intended outcome. | Point of stability
For myopes > 7 D spherical equivalent (SE), a minimum of 75% of eyes should have an uncorrected visual acuity of 20/40 or better at the postoperative interval at which stability has been established. | Point of stability
95% of eyes should have a change of < 1.00 D in manifest refraction spherical equivalent (MRSE) between 2 refractions performed at least 3 months apart, and the mean rate of MRSE change per month should be < 0.04 D. | Point of stability
Distance BSCVA of worse than 20/40 at the postoperative interval at which stability has been established should occur in less than 1% of eyes that had a BSCVA of 20/20 or better before surgery. | Point of stability
Loss of more than 2 lines of BSCVA should occur in less than 5% of eyes | Point of stability
Less than 5% of eyes treated for sphere only should have a magnitude of postoperative manifest refractive astigmatism that varies from baseline cylinder by greater than 2.00 D at the postoperative interval at which stability has been established. | Point of stability
Incidence of Adverse Events to occur in less than 1% of eyes | Postopertive visits

SECONDARY OUTCOMES:
Subject Satisfaction: As measured by a subjective questionnaire, and will be considered as a secondary efficacy variable. | Postoperative visits 3, 6, 9 and 12 months
Incidence of Complications | Postoperative visits
Patient Symptoms: As measured by a subjective questionnaire, will be considered as a secondary safety variable | Preoperative and Postoperative visits 3, 6, 9 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: John Doane, MD, Principal Investigator — Discover Vision Centers; Richard Hoffman, MD, Principal Investigator — Fine, Hoffman, and Packer LLC; Howard Fine, MD, Principal Investigator — Fine, Hoffman, and Packer LLC; Mark Packer, MD, Principal Investigator — FIne, Hoffman, and Packer LLC; David Tanzer, MD, Principal Investigator — US Navy Refractive Surgery Center, San Diego, CA; John Vukich, MD, Principal Investigator — Davis Duehr Dean Eye Clinic; Jon Dishler, MD, Principal Investigator — Dishler Laser Institute
Locations (5):
- United States (5):
  - US Navy Refractive Surgery Center, San Diego, California
  - Dishler Laser Institute, Greenwood Village, Colorado
  - Discover Vision Centers, Kansas City, Missouri
  - Fine, Hoffman, and Packer, Eugene, Oregon
  - Davis Duehr Dean Eye Clinic, Madison, Wisconsin